CLINICAL TRIAL: NCT06744296
Title: Measurable Residual Disease Detection Using Tumor-Informed ctDNA Surveillance After Curative-Intent Treatment in HPV-Independent Squamous Cell Carcinoma of the Head and Neck
Acronym: MRD-DUCHESS
Status: Recruiting | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Haystack Oncology, Inc. (Unknown)
Responsible Party: Principal Investigator, Daniel L. Faden, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2024P002675
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples and tissue ffpe samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Receiving only Surgery: Patients in this group will only be those who receive surgery, and does not receive radiographic testing or chemotherapy.
  Interventions: Other: Blood Draws and Tissue Sample(s)
- Patients receiving chemoradiotherapy: * Newly diagnosed AJCC 8th edition Stage III-IVB mucosal SCC of the head and neck, which includes tumors arising from the oral cavity, nasal cavity, paranasal sinuses, nasopharynx, oropharynx, hypopharynx, and larynx.
  * Available tissue for tumor-informed ctDNA panel creation.
  * Definitive treatment with standard of care surgery (arm 1) or chemoradiotherapy (arm 2)
  Interventions: Other: Blood Draws and Tissue Sample(s)

INTERVENTIONS:
Other: Blood Draws and Tissue Sample(s) — All participants on the study, regardless of arm, will be getting blood draws, and tissue samples.

SUMMARY:
This study will test the ability of a personalized blood test to determine which head and neck cancer patients will have a recurrence after treatment.

DETAILED DESCRIPTION:
This is a two-arm, prospective, observational study of patients with human papillomavirus (HPV)-independent head and neck squamous cell carcinoma (HNSCC) who are receiving curative-intent treatment. Arm 1 will consist of patients who undergo surgery. Arm 2 will consist of patients who undergo chemoradiotherapy.

The study will test the following hypotheses:

1. That applying a tumor-informed minimal residual disease (MRD) assay after completion of curative-intent treatment will accurately discriminate between patients who will eventually experience recurrence (those are MRD positive) and patients who will remain disease-free (those who are MRD negative). The hypothesis is that patients who have detectable ctDNA following treatment-MRD positive patients-will experience recurrent disease within 2 years, while patients who have no detectable ctDNA-MRD negative patients-will remain disease free at 2 years.
2. That measuring MRD after completion of curative-intent treatment will provide a lead time from detectable to clinical diagnosis of recurrent disease of at least 3 months.

The primary outcome is 2-year DFS in patients with detectable vs no detectable ctDNA two weeks after treatment completion.

The study will accrue 75 patients, who will be followed for a minimum of 2 years.

Subjects will have blood draws before, during and following treatment at regular intervals for testing with the assay (Haystack MRD™)

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AJCC 8th edition Stage III-IVB mucosal SCC of the head and neck, which includes tumors arising from the oral cavity, nasal cavity, paranasal sinuses, nasopharynx, oropharynx, hypopharynx, and larynx.
* Available tissue for tumor-informed ctDNA panel creation.
* Definitive treatment with standard of care surgery or chemoradiotherapy is planned to be administered at Massachusetts Eye and Ear Institute (MEEI) or within the Massachusetts General Hospital (MGH) Cancer Center (including but not limited to the Boston, Danvers, and Newton-Wellesley locations).

Exclusion Criteria:

* Patients <18 years of age
* Patients receiving non-standard of care therapy as determined by the clinical investigator
* Participants who have undergone prior surgical resection, excisional biopsy, radiation, and/or chemotherapy for the treatment of HNSCC. Prior incisional biopsies are permitted. Discrepant cases will be reviewed by study PI.
* Participants who are receiving any investigational agents at the time of enrollment.
* Participants with AJCC Stage IVC HNSCC, which includes patients with biopsy-confirmed distant metastatic HNSCC, including but not limited to metastatic spread to the lungs, bones, or liver.
* Active non-HNSCC malignancy.
* Active pregnancy during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage III-IVB mucosal squamous cell carcinoma of the head and neck
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2029-01-06 (Estimated)

PRIMARY OUTCOMES:
2 Years - Disease Free Survival (DFS) | 2 weeks after treatment completion
  2-year disease-free survival (DFS) in patients with detectable vs no detectable ctDNA two weeks after treatment completion

SECONDARY OUTCOMES:
2 Years - Overall Survival (OS) | 2 weeks after treatment completion
  2-year overall survival (OS) in patients with detectable vs no detectable ctDNA two weeks after treatment completion
2 Years - Disease Free Survival (DFS) and Overall Survival (OS) | 4 weeks after treatment completion
  2-year disease-free survival (DFS) and overall survival (OS) in patients with detectable vs no detectable ctDNA four weeks after treatment completion
2 - Years Disease Free Survival (DFS) and Overall Survival (OS) | 6 week after treatment completion
  2-year disease-free survival (DFS) and overall survival (OS) in patients with detectable vs no detectable ctDNA six weeks after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Faden, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States